CLINICAL TRIAL: NCT02198274
Title: A Phase II Uncontrolled Sudy to Evaluate the Antitumour Activity and Safety of Intravenous BIBH 1, Administered in a Weekly Dose of 100 mg in 12 Weeks, in Patients With Metastatic Colorectal Cancer
Brief Title: Intravenous BIBH 1 in Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1152.10
Record Dates: First submitted 2014-07-22; First posted 2014-07-23 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — sibrotuzumab

ARMS (1):
- BIBH 1 (Experimental)
  Interventions: Drug: BIBH 1

INTERVENTIONS:
Drug: BIBH 1 — 100 mg/week
  Other Names: Sibrotuzumab

SUMMARY:
Study to evaluate the anti-tumour activity, safety and pharmacokinetics of unlabelled sibrotuzumab administered weekly (seven days +/- one day) at a dose of 100 mg (a total of 12 administrations) in patients with metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic colorectal cancer International Union Against Cancer (UICC) Stage IV who are progressive under at least two previous chemotherapy regimes or who refused conventional treatment or who are not eligible for conventional treatment
* Progressive disease documented by subsequent computed tomography (CT) or magnetic resonance imaging (MRI) scanning prior to study entry. The last CT or MRI scans must be performed within 1 month before study entry. The first CT or MRI scan should be conducted within 6 months before study entry
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
* Expected survival of ≥ 6 months
* Greater than or equal to 18 years of age
* Platelet count ≥ 100 x 10**9/L
* Total leukocytes ≥ 2500/mm**3
* Alanine aminotransferase/Aspartate aminotransferase (ALT/AST) ≤ 4 x upper limit of normal
* Total bilirubin ≤ 2.0 mg/dl (or 34µmol/L, Systeme International (SI) unit equivalent)
* Serum creatinine ≤ 2.0 mg/dl (0.20 mmol/l)
* Written informed consent in accordance with Good Clinical Practice and local legislation

Exclusion Criteria:

* Active metastatic disease to the central nervous system, exhibited by new or enlarging lesions on CT or MRI scan or within 3 months of treatment (i.e., surgery or radiotherapy) for brain metastases
* Exposure to an investigation agent within 30 days prior to the first BIBH 1 infusion
* Patients who are not fully recovered from surgery (incomplete healing)
* Chemotherapy or immunotherapy within 30 days prior to the first BIBH 1 infusion
* Radiation therapy to the symptomatic sites included for tumour measurements within 30 days prior to study entry
* Previous administration of a murine, chimeric or humanised measurement and/or antibody fragment (e.g. BIBH 1, Panorex)
* Serious illness: e.g., active infections requiring antibiotics, bleeding disorders, patients with known untreated or unstable coronary heart disease (e.g. unstable angina or myocardial infarction within 6 months prior to study entry) or diseases considered by the investigator to have potential for interfering with obtaining accurate results from this study
* Women who are breast-feeding or pregnant
* Men and women of childbearing potential who are unwilling to utilise a medically acceptable method of contraception
* Patients who suffer from autoimmune diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2000-02; Primary Completion 2000-10 (Actual)

PRIMARY OUTCOMES:
Anti-tumour response | 4 weeks after the last administration

SECONDARY OUTCOMES:
Time to tumour progression | up to 16 weeks
Time to loss of response | up to 16 weeks
Disease progression-free survival time | up to 16 weeks
Changes in titers of human anti-human antibody (HAHA) | up to 16 weeks
Incidence and intensity of adverse events graded by Common toxicity criteria (CTC) | up to 16 weeks
Assessment of the maximum toxicity grade observed for each patient | up to 16 weeks
Frequency of on-study deaths | up to 16 weeks
Maximum drug concentration (Cmax) | up to 16 weeks
Minimum drug concentration (Cmin) | up to 16 weeks
Area under the concentration-time curve (AUC) | up to 16 weeks
Total serum clearance (CL) | up to 16 weeks
Volume of distribution at steady state (Vss) | up to 16 weeks
Terminal half-life (t1/2) | up to 16 weeks
Mean residence time (MRT) | up to 16 weeks